CLINICAL TRIAL: NCT00773695
Title: A Multicenter, Randomized, Phase II Clinical Trial to Evaluate the Effect of Avastin in Combination With Neoadjuvant Treatment Regimens on the Molecular and Metabolic Characteristics and Changes in the Primary Tumors With Reference to the Obtained Responses in Patients With Large Primary HER2 Negative Breast Cancers
Brief Title: A Study of Bevacizumab (Avastin) in Combination With Neoadjuvant Treatment Regimens in Participants With Primary Human Epidermal Growth Factor Receptor 2 (HER2) Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Norwegian Radium Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21744
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Aromatase Inhibitors; Bevacizumab; Epirubicin; Fluorouracil; Cyclophosphamide; Paclitaxel; Docetaxel

ARMS (4):
- Chemotherapy (Active Comparator): Participants will receive epirubicine, 5-fluorouracil, and cyclophosphamide (FEC 100) for 12 weeks followed by taxane therapy (paclitaxel or docetaxel) for next 12 weeks.
  Interventions: Drug: Epirubicine; Drug: 5-Fluorouracil (5FU); Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Docetaxel
- Chemotherapy and Bevacizumab (Experimental): Participants will receive epirubicine, 5-fluorouracil, and cyclophosphamide (FEC 100) for 12 weeks followed by taxane therapy (paclitaxel or docetaxel) for next 12 weeks. Participants will also receive concurrent treatment with bevacizumab every 3 weeks for 24 weeks.
  Interventions: Drug: Bevacizumab; Drug: Epirubicine; Drug: 5-Fluorouracil (5FU); Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Docetaxel
- Endocrine Therapy (Active Comparator): Participants will receive aromatase inhibitor therapy at discretion of the investigator for a period of 24 weeks.
  Interventions: Drug: Aromatase Inhibitor
- Endocrine Therapy and Bevacizumab (Experimental): Participants will receive aromatase inhibitor therapy at discretion of the investigator and concurrent treatment with bevacizumab for a period of 24 weeks.
  Interventions: Drug: Aromatase Inhibitor; Drug: Bevacizumab

INTERVENTIONS:
Drug: Aromatase Inhibitor — Participants will receive aromatase inhibitor therapy, at a dose per investigator discretion, once daily for 24 weeks.
  Arms: Endocrine Therapy; Endocrine Therapy and Bevacizumab
Drug: Bevacizumab — Bevacizumab will be administered at a dose of 15 mg/kg as IV infusion every 3 weeks (or 10 mg/kg every other week in participants receiving weekly paclitaxel), for 24 weeks.
  Other Names: Avastin
  Arms: Chemotherapy and Bevacizumab; Endocrine Therapy and Bevacizumab
Drug: Epirubicine — Participants will receive epirubicine at a dose of 100 mg/m^2 as IV infusion every 3 weeks for 12 weeks.
  Arms: Chemotherapy; Chemotherapy and Bevacizumab
Drug: 5-Fluorouracil (5FU) — Participants will receive 5FU at a dose of 600 mg/m^2 as IV infusion every 3 weeks for 12 weeks.
  Arms: Chemotherapy; Chemotherapy and Bevacizumab
Drug: Cyclophosphamide — Participants will receive cyclophosphamide at a dose of 600 mg/m^2 as IV infusion every 3 weeks for 12 weeks.
  Arms: Chemotherapy; Chemotherapy and Bevacizumab
Drug: Paclitaxel — Participants will receive paclitaxel at a dose of 80 mg/m^2 as IV infusion every week for 12 weeks.
  Arms: Chemotherapy; Chemotherapy and Bevacizumab
Drug: Docetaxel — Participants will receive docetaxel at a dose of 100 mg/m^2 as IV infusion every 3 weeks for 12 weeks.
  Arms: Chemotherapy; Chemotherapy and Bevacizumab

SUMMARY:
This study will evaluate the effect of bevacizumab in combination with chemotherapy or endocrine therapy, as preoperative treatment, in participants with HER2 negative breast cancer. Participants will be randomized to receive either chemotherapy (FEC100: Epirubicine 100 milligrams per square meter [mg/m^2], 5-fluorouracil 600 mg/m^2, and cyclophosphamide 600 mg/m^2] for 12 weeks followed by taxane (paclitaxel/docetaxel) for 12 weeks or endocrine therapy (an aromatase inhibitor] daily for 24 weeks) with or without bevacizumab (15 milligrams per kilogram [mg/kg] as intravenous [IV] infusion every 3 weeks up 24 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, HER2-negative, men or pre- or post-menopausal women with primary operable adenocarcinoma of the breast, greater than or equal to (>=) 2.5 centimeters (cm) in size
* Eastern Cooperative Oncology Group (ECOG)/world health organization (WHO) performance status less than or equal to (</=) 2
* Normal baseline cardiac function (Left Ventricular Ejection Fraction [LVEF])

Exclusion Criteria:

* Stage IV (metastatic) disease
* Previous treatment for localized breast cancer less than (<) 24 months from diagnosis of present breast cancer
* Other previous or current cancer except for basal cell cancer or in situ cervical cancer
* Current or recent use of aspirin (greater than [>] 325 milligrams per day)
* Clinically significant cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-11-07 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Messenger Ribonucleic Acid (mRNA) Markers of Pathological Complete Response, as Assessed by Magnetic Resonance Imaging (MRI) | Baseline up to end of study treatment (approximately 24 weeks)

SECONDARY OUTCOMES:
Percentage of Participants With Objective Pathological Complete Response, as Assessed by Clinical Assessment | Baseline up to end of study treatment (approximately 24 weeks)
Percentage of Participants With Type of Surgery | At Surgery (Between Weeks 24 and 25)
  Percentage of participants with different surgery types (for example, Mastectomy, Tumorectomy/Breast conserving therapy (BCT), and Tumorectomy followed by mastectomy) will be reported.
Percentage of Participants With Axillary Lymph Node Dissection Performed | At Surgery (Between Weeks 24 and 25)
Pathological Tumor Size, as Assessed by Histopathological Examination | At Surgery (Between Weeks 24 and 25)
Percentage of Participants With Presence of Tumor Cells Close to Resection Margin | At Surgery (Between Weeks 24 and 25)
Percentage of Participants With Tumor Deposit in Other Body Parts | At Surgery (Between Weeks 24 and 25)
Tumor Free Resection Margin | At Surgery (Between Weeks 24 and 25)
Pathological Tumor Size as Measure Using Caliper | Cycles 1 to 10 (cycle length=21 days), and Week 25
Pathological Tumor Size as Measure Using MRI | Baseline, Weeks 12 and 25
Pathological Tumor Size as Measure Using Mamography | Baseline, Weeks 12 and 25
Pathological Breast Tumor Size as Measure Using Ultrasound | Baseline, Weeks 12 and 25
Pathological Axilla Tumor Size as Measure Using Ultrasound | Baseline, Weeks 12 and 25
Percentage of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status | Screening, Cycles 1 to 10 (cycle length=21 days), and Week 25
Percentage of Participants With Lymph Node Involvement | Cycles 1 to 10 (cycle length=21 days), and Week 25
Percentage of Participants With Objective Tumor Response, as Assessed Using Response Evaluation Criteria in Solid Tumors (RECIST) | Weeks 12 and 25
Percentage of Participants With New Lesions | Weeks 12 and 25
Percentage of Participants With Molecular Changes in Protein Kinase Expression | Baseline up to end of study treatment (approximately 24 weeks)
Percentage of Participants With Molecular Changes in Messenger Ribonucleic Acid (mRNA)/microRNA(miRNA) | Baseline up to end of study treatment (approximately 24 weeks)
Percentage of Participants With Molecular Changes in Protein Expression | Baseline up to end of study treatment (approximately 24 weeks)
Percentage of Participants With Single Nucleotide Polymorphism (SNP) Profiles Predicting Treatment Response | Baseline up to end of study treatment (approximately 24 weeks)
Percentage of Participants With Treatment-Induced Changes in Tumor Cells as Determined by Number of Disseminated Tumor Cells in Bone Marrow | Baseline up to end of study treatment (approximately 24 weeks)
Percentage of Participants With Treatment-Induced Changes in Tumor Cells as Determined by Number of Circulating Tumor Cells in Peripheral Blood | Baseline up to end of study treatment (approximately 24 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Norway (3):
  - The Norvegian Radium Hospital Montebello; Dept of Oncology, Oslo
  - Ullevael Sykehus; Dept of Oncology, Oslo
  - St. Olavs Hospital; Kreftavdelingen, Trondheim

REFERENCES:
- [Derived] Trnkova L, Burikova M, Soltysova A, Ficek A, Plava J, Cumova A, Rojikova L, Jakic K, Sedlackova E, Tichy B, Bystry V, Busato F, Shen Y, Matuskova M, Kucerova L, Oy GF, Maelandsmo GM, Fleischer T, Tost J, Miklikova S, Cihova M, Buocikova V, Smolkova B. Molecular profiling of chemotherapy-resistant breast cancer reveals DNA methylation remodeling associated with the acquisition of paclitaxel resistance. Drug Resist Updat. 2026 Jan 2;85:101350. doi: 10.1016/j.drup.2026.101350. Online ahead of print. PMID 41529624
- [Derived] Hoglander EK, Nord S, Wedge DC, Lingjaerde OC, Silwal-Pandit L, Gythfeldt HV, Vollan HKM, Fleischer T, Krohn M, Schlitchting E, Borgen E, Garred O, Holmen MM, Wist E, Naume B, Van Loo P, Borresen-Dale AL, Engebraaten O, Kristensen V. Time series analysis of neoadjuvant chemotherapy and bevacizumab-treated breast carcinomas reveals a systemic shift in genomic aberrations. Genome Med. 2018 Nov 29;10(1):92. doi: 10.1186/s13073-018-0601-y. PMID 30497530
- [Derived] Reinertsen KV, Engebraaten O, Loge JH, Cvancarova M, Naume B, Wist E, Edvardsen H, Wille E, Bjoro T, Kiserud CE. Fatigue During and After Breast Cancer Therapy-A Prospective Study. J Pain Symptom Manage. 2017 Mar;53(3):551-560. doi: 10.1016/j.jpainsymman.2016.09.011. Epub 2016 Dec 29. PMID 28042070